CLINICAL TRIAL: NCT03655847
Title: Determination of ED50 and ED95 of Single Bolus Dexmedetomidine in General Anesthesia Patients to Produce Acceptable Hemodynamic Outcomes
Brief Title: Acceptable Hemodynamic Changes in Dexmedetomidine for Single Intravenous Bolus Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LCKY2018-32
Record Dates: First submitted 2018-07-02; First posted 2018-08-31 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Postoperative Complications; Pathologic Processes; Neurocognitive Disorders; Mental Disorders; Dexmedetomidine; Hypnotics and Sedatives; Physiological Effects of Drugs; Analgesics; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Delirium; Postoperative Complications; Pathologic Processes; Neurocognitive Disorders; Mental Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dexmedetomidine (Experimental): Drug: Dexmedetomidine dexmedetomidine, 0.1ug/kg up or down Other Name: precedex
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine was injected intravenously 30 minutes before the end of operation. Single bolus is for more than 1 minute. In the first case, the dosage of dexmedetomidine was 0.1 ug/kg. If the cardiovascular reaction was positive (mean arterial pressure or heart rate was more than 20% before intravenous injection), the dosage of Dexmedetomidine in the next patient decreased by a gradient (0.05ug/kg). If the cardiovascular response was negative, the next patient increased the dose of dexmedetomidine by a gradient (0.1ug/kg); if a patient withdrew from the study, the next patient received the same dose as the patient who withdrew.
  Other Names: see arms

SUMMARY:
Dexmedetomidine（DEX）is a potent and highly selective α 2 adrenergic receptor agonist. It has the pharmacological effects of sedation, hypnosis, analgesia, anti-sympathetic and neuroprotective. Its sedative effect is similar to normal sleep, and easy to wake up. DEX is widely used clinically because of its advantages and acceptable side effects. The best clinical use of DEX is uncertain, including intravenous, intramuscular, oral, intralnasal and sublingual administration. Its clinical recommended use is intravenous load infusion for more than 10 minutes, followed by continuous infusion. However, the clinical recommended usage is inconvenient, time-consuming and other shortcomings, for the growing popularity of daytime surgery, will inevitably affect the operation process and turnover. If a suitable dose range of DEX can be found for a single intravenous injection to achieve clinical efficacy quickly without significant hemodynamic effects, this will improve the patient's postoperative recovery. We will speed up the utilization and turnover of medical resources. The aim of this study was to investigate the optimal dosage of DEX for single intravenous injection.

DETAILED DESCRIPTION:
Patients undergoing thyroidectomy under general anesthesia were treated with routine anesthesia induction and maintenance, and DEX was injected intravenously 30 minutes before the end of operation. Single bolus is for more than 1 minute. In the first case, the dosage of DEX was 0.1 ug/kg. If the cardiovascular reaction was positive (MAP or heart rate was more than 20% before intravenous injection), the dosage of DEX in the next patient decreased by a gradient (0.05ug/kg). If the cardiovascular response was negative, the next patient increased the dose of DEX by a gradient (0.1ug/kg); if a patient withdrew from the study, the next patient received the same dose as the patient who withdrew. There were 8 turning points of cardiovascular reaction and the test was completed. The changes of blood pressure and heart rate per minute in 10min were recorded after single bolus. The dosimetric map of patients with DEX was drawn, and the ED50 and ED95 were calculated by probit probabilistic unit regression (Bills method).

ELIGIBILITY:
Inclusion Criteria:

1. volunteer to participate in the study and sign the informed consent;
2. selective operation of thyroid gland whose anesthesia time is less than 2 hours ;
3. aged 18-55 years;
4. ASA I - II;
5. BMI 18~28kg/m2.

Exclusion Criteria:

1. Mallampati grade Ⅲ or Ⅳ;
2. opening degree < 2.5 cm;
3. taking analgesic or sedative drugs for a long time before operation;
4. a history of arrhythmia, bronchial and cardiovascular diseases, abnormal liver function and so on;
5. allergic to dexmedetomidine, similar active ingredients or excipients;
6. G-6-PD deficiency;
7. a history of use of alpha 2 receptor agonists or antagonists.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-03-23 (Estimated); Study Completion 2020-04-23 (Estimated)

PRIMARY OUTCOMES:
Heart rate(HR) | 10min
  HR changes per minutes in 10 minutes after single injection of DEX

SECONDARY OUTCOMES:
Duration of operation | intraoperative, from the beginning of the cut to the end of the seam
  Duration of operation
Anaesthesia time | intraoperative, from initiation of anesthesia induction to cessation of anesthetic use
  Anaesthesia time
Recovery time of anesthesia | within 24 hours
  Recovery time of anesthesia
Mean arterial pressure(MAP) | 10min
  MAP changes per minutes in 10 minutes after single injection of DEX

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, Study Director — The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study complettion.
Access Criteria: Data access request will be reviewed by an external independent review panel.Requestors will be required to sign a Data access agreement.